CLINICAL TRIAL: NCT05357807
Title: Extending and Banding the Roux-en-Y Gastric Bypass
Acronym: UPGRADE
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rijnstate Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NL62168.091.17
Record Dates: First submitted 2021-05-25; First posted 2022-05-03 (Actual); Last update posted 2024-06-21 (Actual); Status verified 2024-06

CONDITIONS: Morbid Obesity
MeSH Terms: conditions — Obesity, Morbid

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Standard RYGB (Active Comparator): 127 patients undergo a standard Roux-en-Y gastric bypass
  Interventions: Procedure: Standard RYGB
- Extended Pouch RYGB (Experimental): 127 patients undergo a Roux-en-Y gastric bypass with an extended pouch.
  Interventions: Procedure: Extended Pouch RYGB
- Banded Extended RYGB (Experimental): 127 patients undergo a Roux-en-Y gastric bypass with a minimizer around the extended pouch.
  Interventions: Procedure: Banded extended pouch RYGB

INTERVENTIONS:
Procedure: Standard RYGB — Roux-en-Y Gastric bypass
  Other Names: S-RYGB
  Arms: Standard RYGB
Procedure: Extended Pouch RYGB — Roux-en-Y gastric bypass with an extended pouch
  Other Names: EP-RYGB
  Arms: Extended Pouch RYGB
Procedure: Banded extended pouch RYGB — Roux-en-Y gastric bypass with a banded extended pouch
  Other Names: BEP-RYGB
  Arms: Banded Extended RYGB

SUMMARY:
The Roux-en-Y gastric bypass (RYGB) has proven to be an effective treatment for morbid obesity by reducing weight and comorbidities. Extending the pouch may improve weightloss without the increase of complications. Some patients regain weight after initially good weightloss. Placing a minimizer around the pouch may prevent weight regain.

DETAILED DESCRIPTION:
The Roux-en-Y gastric bypass (RYGB) has proven to be an effective treatment for morbid obesity by reducing weight and comorbidities. Extending the pouch may improve weightloss without the increase of complications. Some patients regain weight after initially good weightloss. Placing a minimizer around the pouch may prevent weight regain.

A prospective randomize controlled trial.

Study population: alle patients undergoing RYGB are eligible for the study. inclusion criteria are BMI 35-40 kg/m2 with one or more obesity related comorbidities, or BMI > 40 kg/m2 without any comorbidities.

Intervention: Standard RYGB versus an extended pouch RYGB vs a banded-extended RYGB.

ELIGIBILITY:
Inclusion Criteria:

* All patients who are eligible for a primary RYGB

Exclusion Criteria:

* Bariatric surgery in medical history
* Patients with a language barrier which may affect the compliance with medical advice
* Patients with a disease not related to morbid obesity, such as Cushing or drug related.
* Chronic bowel disease for example Crohn's disease or colitis Colitis.
* Renal impairment (MDRD <30)
* Hepatic dysfunction (liver function twice the normal values)
* Pregnancy during follow-up
* Patients with treatment-resistant reflux symptoms.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 375 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2023-06-01 (Actual); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Percentage Total Body Weight Loss (%TBWL) | 3 years
  ((preoperative weight - current weight) / (preoperative weight)) x 100%. Weight loss measured in kilograms

SECONDARY OUTCOMES:
Percentage Excess Weight Loss (%EWL) | 3 years
  ((Preoperative weight - current weight) / (preoperative weight - ideal weight at BMI 25)) x 100%. Weight loss measured in kilograms
BODY-Q: Quality of life after bariatric surgery | 3 years
  BODY-Q: Patient reporterd outcome measurement, The questionnaire measures three domains; health related quality of life, appearance and experience of healthcare. Each domain is composed of independently functioning scales. Each scale contains different statements, which can be scored on four levels ranging from totally disagree to totally agree or from never to always. The sum of levels ranging from 1 to 4 is the raw score of the different scales. This score can be converted into a Rasch Transformed score ranging from 0, worst score, to 100, best score.
BAROS: Quality of life after bariatric surgery | 3 years
  BAROS; evaluates the results of obesity treatments by analyzing 3 domains: weight loss, changes in co-morbidities, and quality of life. Up to 3 points are allowed for each, and points are deducted for complications and reoperations. The final score classifies the results in 5 outcome groups, providing an objective definition of success or failure.
SF-36: Quality of life after bariatric surgery | 3 years
  SF-36; consists of eight scaled scores, which are the weighted sums of the questions in their section. Each scale is directly transformed into a 0-100 scale on the assumption that each question carries equal weight. The lower the score the more disability. The higher the score the less disability
Gastroesophageal reflux disease | 3 years
  GERD-HRQL questionnaire, a higher score on the questionnaire indicates more complaints of gastroesophageal reflux disease.
Change in comorbidities in patients pre- and postoperative | 3 years
  Measuring reduction of diabetes, hypertension, dyslipidemia, osteoarticular disease, OSA

CONTACTS AND LOCATIONS:
Locations (3):
- Netherlands (3):
  - Rijnstate Hospital, Arnhem, Gelderland
  - St. Antonius Ziekenhuis, Nieuwegein, Utrecht
  - NOK West, The Hague

IPD SHARING:
Plan to Share IPD: Undecided